CLINICAL TRIAL: NCT01396005
Title: An Open-Label, One-Period Study in Patients Receiving Methadone or Buprenorphine/Naloxone Maintenance Therapy to Evaluate the Effect of SCH 503034 (Boceprevir) on Either Methadone or Buprenorphine/Naloxone Plasma Concentrations (Protocol No. P08123)
Brief Title: A Study to Evaluate the Pharmacokinetic Effect of SCH 503034 (Boceprevir) on Methadone or Buprenorphine/Naloxone Plasma Concentrations (P08123)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P08123
Record Dates: First submitted 2011-06-28; First posted 2011-07-18 (Estimated); Results first posted 2013-03-11 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C | interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; Methadone; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methadone + boceprevir (Experimental): Participants receive standard methadone maintenance therapy (20-150 mg tablets, liquid, or disket, orally, once per day) on Days 1 through 8 + boceprevir (800 mg [4 x 200 mg capsules], orally, every 8 hours) on Days 2 through 7)
  Interventions: Drug: boceprevir; Drug: methadone
- Buprenorphine/naloxone + boceprevir (Experimental): Participants receive standard buprenorphine/naloxone maintenance therapy (8/2-24/6 mg, tablets, sublingual, once per day) on Days 1 through 8 + boceprevir (800 mg [4 x 200 mg capsules], orally, every 8 hours) on Days 2 through 7
  Interventions: Drug: boceprevir; Drug: buprenorphine/naloxone

INTERVENTIONS:
Drug: boceprevir — boceprevir 800 mg (4 x 200 mg capsules), orally, every 8 hours, Day 2 through Day 7
  Other Names: SCH 503034, Victrelis™
Drug: methadone — methadone, 20-150 mg tablets, liquid, or disket, orally, once per day, Day 1 through Day 8
  Arms: Methadone + boceprevir
Drug: buprenorphine/naloxone — buprenorphine/naloxone 8/2-24/6 mg, tablets, sublingual, once per day, Day 1 through Day 8
  Arms: Buprenorphine/naloxone + boceprevir

SUMMARY:
In this study, participants on methadone or buprenorphine/naloxone maintenance therapy will be given boceprevir. Blood samples will be taken at specified intervals to find out whether boceprevir affects the pharmacokinetics of methadone, buprenorphine, or naloxone.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 18 and 36, inclusive
* Reliable participation in a methadone maintenance or buprenorphine maintenance or buprenorphine/naloxone maintenance program for at least two (2) months prior to Day 1.
* Is receiving once daily oral dose of methadone therapy at a stable

individualized dose for at least 4 weeks, receiving once

daily buprenorphine dose at a stable individualized dose for at 4 weeks with, if on buprenorphine only therapy, naloxone added for at least 2 weeks prior to Day 1.

* 12-lead electrocardiogram (ECG) conduction intervals within gender-specific normal range
* Vital signs within normal range
* Clinical laboratory tests within normal range
* Women who are postmenopausal, surgically sterilized, or premenopausal and use a medically-accepted method of contraception.

Exclusion Criteria:

* Pregnancy, breast feeding, or intention to become pregnant or father a child while on study or within 3 months after end of trial
* History or presence of inflammatory bowel disease, ulcers, or gastrointestinal or rectal bleeding
* History of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection
* History of pancreatic injury or pancreatitis
* History or presence of liver disease or liver injury
* History or presence of impaired renal function
* History of urinary obstruction or difficulty in voiding
* History of any infectious disease within 4 weeks prior to drug administration that in the opinion of the investigator, affects the subject's ability to participate in the trial
* Positive for hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus (HIV)
* Positive screen for drugs with a high potential for abuse such as cocaine, amphetamines, methylenedioxymethamphetamine (MDMA), barbiturates, benzodiazepines, or opiates/opioids
* Excessive use of alcohol in the 2 weeks prior to Day -1, defined as greater than 3 glasses of alcoholic beverages (1 is approximately equivalent to: beer [284 mL/10 oz], wine

  [125 mL/4 oz], or distilled spirits [25 mL/1 oz]) per day.
* Blood donation in the past 60 days
* Previous administration of SCH 503034 (boceprevir)
* Current participation in another clinical study or participation in a clinical study (e.g., laboratory or clinical evaluation) within 30 days of baseline
* Study staff personnel or family members of the study staff personnel
* Demonstrated allergic reactions (eg, food, drug, atopic reactions or asthmatic episodes) that, in the opinion of the investigator and sponsor, interfere with their ability to participate in the trial
* History of malignancy within 5 years from Screening
* Consumption of excessive amounts (equivalent to > 6 cups of brewed coffee/day) of coffee, tea, cola or other caffeinated beverages
* Receipt of any of the following more recently than the washout period prior to Baseline: inhibitors or inducers of cytochrome (CYP) P450, CYP2B6, CYP3A4, and CYP2D6; or oral contraceptives containing drospirenone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Hulskotte EG, Bruce RD, Feng HP, Webster LR, Xuan F, Lin WH, O'Mara E, Wagner JA, Butterton JR. Pharmacokinetic interaction between HCV protease inhibitor boceprevir and methadone or buprenorphine in subjects on stable maintenance therapy. Eur J Clin Pharmacol. 2015 Mar;71(3):303-11. doi: 10.1007/s00228-014-1789-4. Epub 2015 Feb 11. PMID 25666027

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Methadone + Boceprevir | Buprenorphine/Naloxone + Boceprevir
Started | 10 | 11
Completed | 10 | 9
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Non-compliance with protocol | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methadone + Boceprevir | Buprenorphine/Naloxone + Boceprevir | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.2 (10.2) | 33.2 (29.0) | 33.7 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration Versus Time Curve (AUC) at Steady State of Methadone Enantiomers When Administered With or Without Boceprevir
Description: AUC is a measure of the amount of drug in the blood over time, measured at steady state (time at which the amount of drug eliminated by the body is in equilibrium with the amount taken in). The Day 1, 0 through 24 hour samples were for methadone levels in the absence of boceprevir co-administration. The Day 7, 0 through 24 hour samples were for methadone levels in the presence of boceprevir co-administration. The Day 5 and 6 predose samples were to check steady state for methadone + boceprevir.
Time Frame: Methadone samples collected Day 1, 0 (predose) through 24 hours post-dose (Day 2). Boceprevir and methadone samples collected Day 7, 0 (predose) through 24 hours post-dose (Day 8). Predose samples also collected on Days 5-6.
Population: All participants receiving standard methadone maintenance therapy + boceprevir
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng.hr/mL)/mg
Groups:
- Methadone Alone; Methadone + Boceprevir: Participants receive standard methadone maintenance therapy (20-150 mg tablets, liquid, or disket, orally, once per day) on Days 1 through 8 + boceprevir (800 mg [4 x 200 mg capsules], orally, every 8 hours) on Days 2 through 7)
Arm/Group | Methadone Alone | Methadone + Boceprevir
Number analyzed (Participants) | 10 | 10
(ng.hr/mL)/mg
  R-methadone | 50.1 (29) | 42.4 (23)
  S-methadone | 56.9 (52) | 44.6 (43)

2. Primary Outcome: Maximum Concentration (Cmax) at Steady State of Methadone Enantiomers When Administered With or Without Boceprevir
Description: Cmax is a measure of the maximum level of drug in the blood, measured at steady state (time at which the amount of drug eliminated by the body is in equilibrium with the amount taken in). The Day 1, 0 through 24 hour samples were for methadone levels in the absence of boceprevir co-administration. The Day 7, 0 through 24 hour samples were for methadone levels in the presence of boceprevir co-administration. The Day 5 and 6 predose samples were to check steady state for methadone + boceprevir.
Time Frame: as for outcome 1
Population: All participants receiving standard methadone maintenance therapy + boceprevir
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng/mL)/mg
Arm/Group | Methadone Alone | Methadone + Boceprevir
Number analyzed (Participants) | 10 | 10
(ng/mL)/mg
  R-methadone | 2.94 (22) | 2.63 (59)
  S-methadone | 3.69 (39) | 3.07 (69)

3. Primary Outcome: AUC of Buprenorphine (Administered in Combination With Naloxone) at Steady State With or Without Boceprevir
Description: AUC is a measure of the amount of drug in the blood over time, measured at steady state (time at which the amount of drug eliminated by the body is in equilibrium with the amount taken in). The Day 1, 0 through 24 hour samples were for buprenorphine/naloxone levels in the absence of boceprevir co-administration. The Day 7, 0 through 24 hour samples were for buprenorphine/naloxone levels in the presence of boceprevir co-administration. The Day 5 and 6 predose samples were to check steady state for buprenorphine/naloxone + boceprevir.
Time Frame: Buprenorphine/naloxone samples collected Day 1, 0 (predose) through 24 hours post-dose (Day 2). Boceprevir and buprenorphine/naloxone samples collected Day 7, 0 (predose) through 24 hours post-dose (Day 8). Predose samples also collected on Days 5-6.
Population: All participants on Day 1; 2 participants were discontinued from study (Days 2-8).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (pg.hr/mL)/mg
Groups:
- Buprenorphine/Naloxone Alone; Buprenorphine/Naloxone + Boceprevir: Participants receive standard buprenorphine/naloxone maintenance therapy (8/2-24/6 mg, tablets, sublingual, once per day) on Days 1 through 8 + boceprevir (800 mg [4 x 200 mg capsules], orally, every 8 hours) on Days 2 through 7
Arm/Group | Buprenorphine/Naloxone Alone | Buprenorphine/Naloxone + Boceprevir
Number analyzed (Participants) | 11 | 9
(pg.hr/mL)/mg | 3020 (55) | 4040 (43)

4. Primary Outcome: Cmax of Buprenorphine (Administered in Combination With Naloxone) at Steady State With or Without Boceprevir
Description: Cmax is a measure of the maximum level of drug in the blood, measured at steady state (time at which the amount of drug eliminated by the body is in equilibrium with the amount taken in). The Day 1, 0 through 24 hour samples were for buprenorphine/naloxone levels in the absence of boceprevir co-administration. The Day 7, 0 through 24 hour samples were for buprenorphine/naloxone levels in the presence of boceprevir co-administration. The Day 5 and 6 predose samples were to check steady state for buprenorphine/naloxone + boceprevir.
Time Frame: as for outcome 3
Population: All participants on Day 1; 1 participant discontinued from study on Day 6.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (pg/mL)/mg
Arm/Group | Buprenorphine/Naloxone Alone | Buprenorphine/Naloxone + Boceprevir
Number analyzed (Participants) | 11 | 10
(pg/mL)/mg | 440 (52) | 545 (45)

5. Secondary Outcome: AUC of Naloxone (Administered in Combination With Buprenorphine) at Steady State With or Without Boceprevir
Description: as for outcome 3
Time Frame: as for outcome 3
Population: All participants on Day 1; 2 participants were discontinued from study (Days 2-8).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (pg.hr/mL)/mg
Arm/Group | Buprenorphine/Naloxone Alone | Buprenorphine/Naloxone + Boceprevir
Number analyzed (Participants) | 11 | 9
(pg.hr/mL)/mg | 157 (62) | 224 (56)

6. Secondary Outcome: Cmax of Naloxone (Administered in Combination With Buprenorphine) at Steady State With or Without Boceprevir
Description: as for outcome 4
Time Frame: as for outcome 3
Population: All participants on Day 1; 1 participant discontinued on Day 6.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (pg/mL)/mg
Arm/Group | Buprenorphine/Naloxone Alone | Buprenorphine/Naloxone + Boceprevir
Number analyzed (Participants) | 11 | 10
(pg/mL)/mg | 58.5 (87) | 65.2 (70)

ADVERSE EVENTS:
Arm/Group | Methadone + Boceprevir | Buprenorphine/Naloxone + Boceprevir
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 10/10 | 9/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methadone + Boceprevir (N=10) | Buprenorphine/Naloxone + Boceprevir (N=11)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (3)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Product taste abnormal (General disorders) | 2 (2) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 5 (5)
Headache (Nervous system disorders) | 3 (4) | 3 (4)
Somnolence (Nervous system disorders) | 3 (3) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 2 (2)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus generalized (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the Sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication (including, without limitation, slides and texts of oral or other public presentations and texts of any transmission through any electronic media, eg, any computer access system such as the Internet, World Wide Web, etc) that report any results of the trial.